CLINICAL TRIAL: NCT03290209
Title: Randomized Controlled Trials Comparing Clinical Outcomes of Laparoscopic D1 Versus D2 Lymphadenectomy for Elderly Patients With Advanced Gastric Cancer
Brief Title: Clinical Outcomes of Laparoscopic D1 Versus D2 Lymphadenectomy for Elderly Patients With Advanced Gastric Cancer
Acronym: D1D2
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Chang-Ming Huang, Prof., Director, Head of gastric surgery, Principal Investigator, Clinical Professor, Fujian Medical University Union Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-03
Record Dates: First submitted 2017-09-19; First posted 2017-09-21 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Stomach Neoplasm
Keywords: Stomach Neoplasm; Elderly Patients; Laparoscopic D1 Lymphadenectomy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic D1 Lymphadenectomy (Experimental): Laparoscopic D1 Lymphadenectomy will be performed for the treatment of patients assigned to this group.
  Interventions: Procedure: Laparoscopic D1 Lymphadenectomy
- Laparoscopic D2 Lymphadenectomy (Active Comparator): Laparoscopic D2 Lymphadenectomy will be performed for the treatment of patients assigned to this group.
  Interventions: Procedure: Laparoscopic D2 Lymphadenectomy

INTERVENTIONS:
Procedure: Laparoscopic D1 Lymphadenectomy — After exclusion of T4b, bulky lymph nodes, or distant metastasis case, laparoscopic D1 Lymphadenectomy will be performed in the experimental group.
  Arms: Laparoscopic D1 Lymphadenectomy
Procedure: Laparoscopic D2 Lymphadenectomy — After exclusion of T4b, bulky lymph nodes, or distant metastasis case, laparoscopic D2 Lymphadenectomy will be performed in the comparator group.
  Arms: Laparoscopic D2 Lymphadenectomy

SUMMARY:
The purpose of this study is to explore the clinical outcomes of laparoscopic D1 lymphadenectomy for elderly patients with advanced gastric adenocarcinoma（cT2-4a, N-/+, M0）

DETAILED DESCRIPTION:
Gastrectomy with D2 lymphadenectomy is considered the gold standard treatment for advanced gastric cancer. However, some studies show that age or comorbidities is the relevant predictor of postoperative complications, conditioning the safety of the surgical procedure itself, thus affect the survial. Even with the advances in surgical techniques and care, age still is a significant risk for postoperative morbidity and mortality. Therefore, elderly patients with gastric cancer could receive minimally invasive surgery with reduced nodal dissection, i.e., D1 lymphadenectomy, in order to prevent postoperative complications. Laparoscopic surgery is a minimally invasive operation and is proved to be an acceptable alternative to open surgery. At present, there is no RCTs to confirm the safety and effectiveness of laparoscopic D1 lymphadenectomy for elderly patients with advanced gastric adenocarcinoma. This study is to compare the clinical outcomes of laparoscopic D1 versus D2 lymphadenectomy for elderly patients with advanced gastric adenocarcinoma（cT2-4a, N-/+, M0）to evaluate the safety of laparoscopic D1 lymphadenectomy, and to verify its results in terms of survival in elderly patients with advanced gastric adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age over or equal to 75 years
2. Primary gastric adenocarcinoma (papillary, tubular, mucinous, signet ring cell, or poorly differentiated) confirmed pathologically by endoscopic biopsy, including gastric multiple primary carcinoma
3. cT2-4a(clinical stage tumor), N-/+, M0 at preoperative evaluation according to the American Joint Committee on Cancer (AJCC) Cancer Staging Manual 8th Edition
4. expected to perform distal, total or proximal gastrectomy to obtain R0 resection sugicall results.
5. Performance status of 0 or 1 on ECOG (Eastern Cooperative Oncology Group) scale
6. ASA (American Society of Anesthesiology) class I to III
7. Written informed consent

Exclusion Criteria:

1. Severe mental disorder
2. History of previous upper abdominal surgery (except laparoscopic cholecystectomy)
3. History of previous gastric surgery (including ESD/EMR (Endoscopic Submucosal Dissection/Endoscopic Mucosal Resection )for gastric cancer)
4. Enlarged or bulky regional lymph node （diameter over 3cm）supported by preoperative imaging
5. History of other malignant disease within the past 5 years
6. History of previous neoadjuvant chemotherapy or radiotherapy
7. History of unstable angina or myocardial infarction within the past 6 months
8. History of cerebrovascular accident within the past 6 months
9. History of continuous systematic administration of corticosteroids within 1 month
10. Requirement of simultaneous surgery for other disease
11. Emergency surgery due to complication (bleeding, obstruction or perforation) caused by gastric cancer
12. FEV1<50% of the predicted values

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
3-year disease specific survival rate | 36 months
  the rate of 3-year disease specific survival

SECONDARY OUTCOMES:
3-year overall survival rate | 36 months
  the rate of 3-year overall survival rate
3-year disease free survival rate | 36 months
  the rate of 3-year disease free survival
number of retrieved lymph nodes | 1 day
  number of retrieved lymph nodes
number of positive lymph nodes | 1 day
  number of positive lymph nodes
intraoperative blood loss | 1 day
  intraoperative blood loss
the rate of conversion to laparotomy | 1 day
  the rate of conversion to laparotomy
overall postoperative morbidity rate | 30 days
  Refers to the incidence of early postoperative complications. The early postoperative complication are defined as the event observed within 30 days after surgery.
overall postoperative mortality rate | 30 days
  the rate of surgical mortality
Time to first ambulation | 30 days
  Time to first ambulation in hours is used to assess the postoperative recovery course.
Time to first flatus | 30 days
  Time to first flatus in days is used to assess the postoperative recovery course.
Time to first liquid diet | 30 days
  Time to first liquid diet in days is used to assess the postoperative recovery course.
Time to first soft diet | 30 days
  Time to first soft diet in days is used to assess the postoperative recovery course.
Duration of postoperative hospital stay | 30 days
  Duration of postoperative hospital stay in days is used to assess the postoperative recovery course.
The variation of white blood cell count | Preoperative 3 days and postoperative 1, 3, and 5 days
  The values of white blood cell count from peripheral blood before operation and on postoperative day 1, 3, 5 are recorded to access the inflammatory and immune response.
The variation of hemoglobin | Preoperative 3 days and postoperative 1, 3, and 5 days
  The values of hemoglobin in gram/liter from peripheral blood before operation and on postoperative day 1, 3, 5 are recorded to access the inflammatory and immune response.
The variation of C-reactive protein | Preoperative 3 days and postoperative 1, 3, and 5 days
  The values of C-reactive protein IN milligram/liter from peripheral blood before operation and on postoperative day 1, 3, 5 are recorded to access the inflammatory and immune response.
The variation of prealbumin | Preoperative 3 days and postoperative 1, 3, and 5 days
  The values of prealbumin in gram/liter from peripheral blood before operation and on postoperative day 1, 3, 5 are recorded to access the inflammatory and immune response.
operation time | 1 day
  operation time

CONTACTS AND LOCATIONS:
Overall Officials: Changming Huang, Professor, Principal Investigator — Fujian Medical University Union Hospital
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China